CLINICAL TRIAL: NCT03169647
Title: Evaluating the Effectiveness of Treatment for Metacognition in Moderate and Severe Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-936-16
Record Dates: First submitted 2017-04-11; First posted 2017-05-30 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): listening-based protocol (type A)
  Interventions: Behavioral: Listening-based intervention
- Control (Placebo Comparator): listening-based protocol (type B)
  Interventions: Behavioral: Listening-based intervention

INTERVENTIONS:
Behavioral: Listening-based intervention — Participants will listen to pre-specified material on a CD

SUMMARY:
Metacognition, in-the-moment awareness of performance while engaging in cognitive tasks, is negatively affected by traumatic brain injury (TBI). Metacognitive deficits can greatly reduce quality of life for individuals with TBI as functioning in this domain has been closely linked with successful independent living and community re-integration. Problematically, there are currently no empirically validated treatment options that address metacognitive deficits after TBI. Recent research in healthy samples demonstrates that specific listening interventions may alter neural activation in brain works associated with metacognition and can improve metacognitive functioning; however, it remains unknown if these effects generalize to individuals with TBI. Thus, the objective of the proposed study is to use a double-blind, placebo controlled randomized clinical trial to determine the efficacy of applying a specific listening intervention to improve metacognition after TBI and to employ functional magnetic resonance imaging (fMRI) to document the neural mechanisms by which the intervention operates.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of moderate or severe brain injury
* between the ages of 18 and 59.
* able to read and speak English fluently.
* TBI at least 1 year ago.

Exclusion Criteria:

* pregnant.
* left-handed.
* color-blind.
* diagnosed with significant psychiatric illness (e.g., bipolar, schizophrenia).
* receiving or have received inpatient and/or rehabilitative treatment for substance use.
* diagnosis of a neurological condition other than TBI (e.g., epilepsy, multiple sclerosis, stroke).
* any metal in my body that has not been declared MRI-safe by my physician.
* impaired independent use of either hand.
* any of the following in/on my body that may interfere with MRI: pacemaker, implanted electrical devices, brain stimulators, particular types of dental implants, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves, and internal hearing aids), permanent eyeliner, implanted delivery pumps, or shrapnel fragments.
* history of engaging in welding and/or metal working activities.
* formal training or am a current practitioner of yoga, meditation, and/or mindfulness.
* currently involved in any other type of thinking skills and/or emotional treatment, such as psychotherapy.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Goodman and Kruskal gamma coefficient on MRI-based metacognitive task | 7 weeks
  While participants are in the scanner, they will perform a metamemory paradigm that involves the completion of 2 components per trial: 1) a memory task (a non-verbal recognition task), and 2) a metacognitive task that immediately follows completion of every recognition item. Accuracy of metacognitive functioning can be quantified using the Goodman and Kruskal gamma coefficient,16 a value between -1 and 1, indicating the discrepancy between the participant's judgment and objective performance that is commonly used in the metacognitive literature.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No